CLINICAL TRIAL: NCT02980042
Title: Evaluating the Tolerability and Safety Profile of Switching From Rituximab to Ocrelizumab: A Real World Evaluation of Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: Safety of Switching From Rituximab to Ocrelizumab in MS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1354
Record Dates: First submitted 2016-11-09; First posted 2016-12-02 (Estimated); Results first posted 2020-01-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Switching Group (Experimental): 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Interventions: Drug: Ocrelizumab
- Comparator Group (Active Comparator): Standard of care rituximab doses are 1000 mg infusion given as first dose followed by 500mg (or 1000 mg if evidence of early B cell recovery) infusion every 6 months thereafter. Rituximab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and rituximab should be infused through a dedicated line
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Ocrelizumab — A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
  Other Names: Ocrevus
  Arms: Switching Group
Drug: Rituximab — A chimeric monoclonal antibody against CD20.
  Other Names: Rituxan
  Arms: Comparator Group

SUMMARY:
This is a prospective between and within group observational study to determine differences in tolerability, immunogenicity and safety related outcomes for 100 multiple sclerosis (MS) patients who have been administered at least two infusions of rituximab, six months apart and are willing to be switched to ocrelizumab compared to a 100 patients who are continuing on rituximab as a comparison cohort from the clinic population treated as part of clinical care.

DETAILED DESCRIPTION:
Studies of rituximab, a chimeric monoclonal antibody against CD20 have shown that B-cell depletion is of clinical beneﬁt as a potential treatment in relapsing forms of multiple sclerosis (MS).1 Ocrelizumab is a humanized monoclonal antibody that targets CD20 and selectively depletes CD20 expressing cells, while preserving the capacity for B cell reconstitution. When compared with rituximab, ocrelizumab is associated with increased antibody-dependent cell-mediated cytotoxic eﬀects, and reduced complement-dependent cytotoxic eﬀects in vitro.2 By increasing antibody-dependent cell mediated cytotoxic eﬀects, ocrelizumab might modulate tissue-dependent mechanisms of pathogenic response more eﬀectively compared to rituximab. As a humanized molecule, ocrelizumab is expected to be less immunogenic with repeated infusions and might thus present a more favorable safety profile when compared to rituximab.2

Despite rituximab's current off label use in the treatment of MS, currently there is only data available from phase 2 trials. The HERMES group conducted a phase 2, double-blind, 48-week trial involving 104 patients with relapsing forms of MS; 69 patients received 1000 mg of intravenous rituximab and 35 patients received placebo on days 1 and 15.3 A significantly higher number of patients in the rituximab group (78.3%) versus the placebo group (40.0%) had an infusion related reaction (IRR) events within 24 hours after the first infusion. Within 24 hours after the second infusion, fewer patients in the rituximab group (20.3%) than in the placebo group (40%) had similar events. A majority of the rituximab group with IRR events (92.6%) were classified as mild to moderate (grade 1 or 2) in severity.

Safety data from the Investigators Brochure on the OPERA I and II phase 3 trials comparing ocrelizumab to interferon β-1a on relapsing MS patients showed that IRRs were the most common adverse events experienced by patients treated with 600 mg of ocrelizumab.4 The percentage of patients experiencing IRRs was higher in the ocrelizumab group (relapsing forms of MS: 34.3%; primary progressive forms of MS 39.9%) compared with the interferon β-1a (active control) group who received placebo infusions (relapsing forms of MS: 9.7%; primary progressive forms of MS: 25.5%). The rate of IRRs was highest during the first infusion or Dose 1 (27.5% on Day 1; 4.71% on Day 15 of Dose 1) and decreased over time (13.7%; 9.6% and 7.8% following Dose 2, 3, and 4 respectively) for the ocrelizumab treated group. Comparatively, interferon β-1a users experienced 6.5% of IRRs on Day 1, 2.58% on Day 15, < 2.00% after doses 2, 3 and 4 respectively. The reported IRRs were primarily mild-to-moderate in severity (Grades 1 and 2). Serious IRRs occurred in 0.1% and 1.0% respectively of relapsing and progressive patients and treated with ocrelizumab.

Clinical data describing the efficacy and tolerability profile of rituximab and ocrelizumab has utilized populations with different prior treatment characteristics. In the phase 2 HERMES trials, a majority (78.5%) of rituximab patients had been previously been treated with a disease modifying therapy in the last 2 years.3 In contrast, the OPERA I and II phase 3 clinical trials, a majority of ocrelizumab patients (72.9% in OPERA I and 73.8% in OPERA II) represented a treatment naïve population.4 Examining IRRs in patients who have switched from rituximab to ocrelizumab versus those continuing on rituximab will examine the magnitude of the IRRs and subsequent tolerability of ocrelizumab in a real world population.

Earlier concepts of MS disease pathology have suggested that pathogenic T cells are sufficient for the full expression of MS. However, it is now evident that full autoimmune B cells and humoral immune mechanisms also play key roles. 5 Ocrelizumab is a humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells. CD20 is a B cell surface molecule that is expressed on pre B cells and mature B cells, but not expressed earlier in the development of B cells or on mature plasma cells. In all three ocrelizumab studies (with relapsing and progressive populations), treatment with 600 mg of ocrelizumab led to rapid and complete depletion of circulating CD19+ B cells within 14 days post treatment. 4 B cell depletion was sustained throughout treatment period. The median time to repletion of B cells was 72 weeks (range 27-175 weeks). We hypothesize that in switching rituximab treated patients to ocrelizumab, the proportion of patients with B cell depletion (< 1%) 6 months after the first and third infusion of ocrelizumab will be the same as the baseline assessment which will be 6 months after the last dose of rituximab and similar to findings in OPERA I and II.

Immunogenicity results from the OPERA I and II trials examined the number of patients who had treatment induced anti-drug antibodies (ADA) to ocrelizumab. 4 Of the 807 patients who received ocrelizumab and had an ADA assay from a post baseline sample during the controlled treatment period, 3 patients (0.4%) showed treatment induced ADA to ocrelizumab. Of these, 1 patient tested positive for neutralizing antibodies (NAB) to ocrelizumab. During the open label extension phase, the prevalence of ADA continued to remain low with post baseline incidence of 1.9% (2/103 with treatment induced ADA). Currently there is little evidence examining the prevalence of treatment induced ADAs to both rituximab and ocrelizumab in patients that switch from the former to the latter in comparison to continuing rituximab patients. Therefore, we will perform assays to detect ADAs to both rituximab and ocrelizumab in all patients switching from rituximab to ocrelizumab at Day 1, 6 months and 12 months on ocrelizumab.

Finally, IRRs have been hypothesized to be a reaction by autoantibodies to the treatment drug or possibly from the release of cytokines from CD20 expressing cells as they are destroyed by ocrelizumab causing a "cytokine storm". Understanding this process may lead to mechanisms that may aid in ameliorating these infusion reactions. If they are associated with ADA, then it might be possible to predictively premedicate these patients only. Alternatively, if they are associated with cytokine release, it may be possible to eliminate premedication in patients who are already CD20+cell depleted in subsequent infusions. Therefore, we will assay the profile of certain cytokines in the serum 4 hours after start of ocrelizumab infusion.

With ocrelizumab expected to enter the MS therapeutic market within the next year, we expect third party payers within and outside the US will require that the FDA or EMA approved versions of anti-CD20 monoclonal antibodies be used in the treatment of MS, namely ocrelizumab. Currently, we estimate several thousand MS patients in the US and Sweden are taking rituximab currently. Thus, it will be important to demonstrate that switching from a chimeric anti-CD20 to a fully humanized anti-CD20 does not lead to unexpected infusion reactions and does not increase the probability of development of anti-drug antibodies.

The Rocky Mountain MS Center (RMMSC) at the University of Colorado Anschutz Medical Campus prescribed rituximab infusions for 533 MS patients in the last 12 months, of which 323 patients received their infusion at the University of Colorado Hospital's Outpatient Infusion Center between September, 2015-March, 2016. The RMMSC is one of the few sites nationwide with large numbers of MS patients treated with rituximab. With the anticipated approval of ocrelizumab, current rituximab users are being counselled by their MS providers at RMMSC to consider switching to ocrelizumab post approval, particularly if US Payers adopt the FDA approved version as the preferred anti-CD20 agent for MS.

ELIGIBILITY:
Inclusion Criteria:

Switching group:

* Current active patient of RMMSC
* 18-65 years
* Diagnosis of relapsing forms of MS
* Completed ≥ two doses of rituximab with the last dose having been administered:

  1. Within 12 months of screening and
  2. At least 6 months prior to the first planned infusion of study drug
* Are receiving their current infusions of rituximab at the University of Colorado Outpatient Infusion Center
* Have discussed the possibility of switching to ocrelizumab with their MS provider
* Screened for Hepatitis B and C and TB within 2 years of first dose of ocrelizumab
* A negative serum pregnancy test must be available for premenopausal women and for women <12 months after the onset of menopause, unless they have undergone surgical sterilization.
* Women of childbearing potential must agree to use a "highly effective", hormonal form of contraception or two "effective" forms of non-hormonal contraception. Contraception must continue for the duration of study treatment and for at least three months after the last dose of study treatment
* Are able to complete patient reported outcomes developed as English written scales.
* Must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with local regulatory requirements

Comparator group:

* Current active patient of RMMSC
* 18-65 years
* Diagnosis of relapsing forms of MS
* Completed ≥ two doses of rituximab with the last dose having been administered within 12 months of screening as standard of care
* Are receiving their current infusions of rituximab as standard of care at the University of Colorado Outpatient Infusion Center and will continue to do so
* Are willing to be followed for up to two additional rituximab infusions during the study period as standard of care
* Must be able and willing to give meaningful, written informed consent prior to participation in the trial, in accordance with local regulatory requirements

Exclusion Criteria:

Both groups:

* Pregnant or lactating women
* Hypersensitivity to trial medications
* Hepatic Dysfunction (liver enzymes are 5 times greater than normal)
* History of Congestive Heart Failure
* Any history of a positive blood assay for Hepatitis B or C
* Any history of TB or a positive Quantiferon Gold Assay
* Concurrent use of immunosuppressant medications
* Any history of immunodeficiency or other medical condition increasing risk of anti-CD 20 therapy.
* No serious infection at the time of a scheduled study infusion.
* Any medical, psychiatric or other condition that could result in the patient not being able to give fully informed consent, or to comply with the protocol requirements as determined by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Vollmer, MD, Principal Investigator — University of Colorado, Denver; Kavita Nair, PhD, Principal Investigator — University of Colorado, Denver; Enrique Alvarez, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switching Group | Comparator Group
Started | 100 | 100
Completed | 93 (All 100 subjects completed their Week 24 infusion. 7 subjects did not complete the 12 month visit.) | 100
Not Completed | 7 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Insurance issues/treatment plan changes | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switching Group | Comparator Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.30 (11.01) | 43.82 (9.97) | 44.56 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 75 | 143
  Male | 32 | 25 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 92 | 89 | 181
  Other | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/African American | 5 | 12 | 17
  White | 90 | 82 | 172
  Asian | 1 | 0 | 1
  Native American | 0 | 1 | 1
  Other | 4 | 5 | 9
Expanded Disability Status Scale (EDSS) [Median (Inter-Quartile Range); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is a tool used to assess disability in multiple sclerosis patients. Scores range from 0 (least disabled) to 10 (most severely disabled) in increments of 0.5. Population: EDSS was not collected for the comparator group at baseline. EDSS is only available for the Switching group.
  units on a scale
    number analyzed (Participants) | 100 | 0 | 100
    (all) | 3.5 [2 to 6] |  | 3.5 [2 to 6]
Patient Determined Disease Steps (PDDS) [Median (Inter-Quartile Range); unit: units on a scale] — The Patient Determined Disease Steps (PDDS) is a patient reported measurement tool used to assess level of disability that the patient perceives in multiple sclerosis patients. Scores range from 0 (least perceived disability) to 10 (most severe perceived disability). Population: PDDS was not collected for the comparator group. PDDS is only available for the Switching group.
  units on a scale
    number analyzed (Participants) | 100 | 0 | 100
    (all) | 3 [1 to 4] |  | 3 [1 to 4]
Disease Duration [Mean (Standard Deviation); unit: years] | 11.20 (7.91) | 11.32 (7.97) | 11.26 (7.92)
Number of Years on rituximab [Mean (Standard Deviation); unit: years] | 2.38 (1.37) | 2.44 (1.45) | 2.41 (1.41)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Infusions With >= 1 IRR Between the Switching and Comparator Groups
Description: The investigators will report the proportion of infusions with >= 1 IRR (infusion-related reaction) between the switching and comparator groups. Data was collected at Day 1, Day 15, and Week 24 and combined to determine the overall proportion of IRRs over the life of the study.
Time Frame: Day 1, Day 15, Week 24
Population: The Switching group received 3 infusions (Day 1, Day 15 and week 24), and the Comparator group received 2 infusions. There were a total of 300 infusions in the Switching group and 200 in the Comparator group. Proportion of IRRs are taken out of total number of infusions.
Measure: Number; unit: percentage of infusions with IRRs
Units Other Than Participants: Infusions
Arm/Group | Switching Group | Comparator Group
Number analyzed (Participants) | 100 | 100
Number analyzed (Infusions) | 300 | 200
percentage of infusions with IRRs | 10 | 14
Statistical Analysis 1: Comparison: Switching Group vs Comparator Group; Test type: Superiority; p = 0.1996, Generalized estimating equations; GEE was necessary because there are repeated measures on subjects; Risk Ratio (RR) = .6616, 95% CI 2-sided [.3666 to 1.1942] — This is comparing the Switching group to the Comparator group

2. Primary Outcome: Difference in the Total Number of IRRs After Each Infusion of Ocrelizumab Compared to Rituximab Infusions in the Comparator Group.
Description: The investigators will report the difference in the total number of IRRs after each infusion of ocrelizumab compared to combined rituximab infusions in the comparator group.
Time Frame: Pre-study (Enrollment), Day 1, Day 15, Week 24
Population: Participants in the comparator group were assessed to have had two pre-study infusions at time of enrollment. A retrospective chart review was conducted to determine the number of IRRs experienced during these previous infusions. The collected number of IRRs was used as a comparison measure against the switching group.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Switching Group | Comparator Group
Number analyzed (Participants) | 100 | 100
Number analyzed (Infusions) | 100 | 200
Infusions
  Pre-study infusions: number analyzed (Participants) | 0 | 100
  Pre-study infusions: number analyzed (Infusions) | 0 | 200
  Pre-study infusions |  | 28
  Day 1: number analyzed (Participants) | 100 | 0
  Day 1: number analyzed (Infusions) | 100 | 0
  Day 1 | 14 |
  Day 15: number analyzed (Participants) | 100 | 0
  Day 15: number analyzed (Infusions) | 100 | 0
  Day 15 | 4 |
  Week 24: number analyzed (Participants) | 100 | 0
  Week 24: number analyzed (Infusions) | 100 | 0
  Week 24 | 12 |
Statistical Analysis 1: Comparison: Switching Group vs Comparator Group; Test type: Superiority; p = 1.0000, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = 1.0000, 95% CI 2-sided [.5299 to 1.8872] — Comparing Switching group Day 1 to combined Comparator group
Statistical Analysis 2: Comparison: Switching Group vs Comparator Group; Test type: Superiority; p = 0.0053, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = .2857, 95% CI 2-sided [.1006 to .8114] — Switching group Day 15 was compared to combined Comparator group
Statistical Analysis 3: Comparison: Switching Group vs Comparator Group; Test type: Superiority; p = 0.6474, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = .8571, 95% CI 2-sided [.4385 to 1.6753]

3. Primary Outcome: Severity of IRRs Following the Day 1 Infusion of Ocrelizumab in the Switching and the Comparator Groups Infusions
Description: The severity of IRRs will be assessed following each infusion of ocrelizumab in the switching and comparator group using the National Cancer Institute's Common Terminology for Adverse Events Scale (Grades range from 1-5, with higher Grades indicating more severe reactions). The frequency of each severity grade of IRR will be compared in a similar fashion .
Time Frame: Day 1, pre-study infusions
Population: The Switching group received 3 infusions (Day 1, Day 15 and week 24), and the Comparator group received 2 infusions prior to enrollment (as assessed via retrospective chart review). This analysis is comparing IRRs of the Switching group's Day 1 infusion, with the comparator group's pre-study infusion 1 and 2.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Switching Group | Comparator Group
Number analyzed (Participants) | 100 | 200
Number analyzed (Infusions) | 100 | 200
Infusions
  No Infusion Reaction | 86 | 172
  Grade 1 Infusion Reaction | 8 | 3
  Grade 2 Infusion Reaction | 6 | 25
  Grade 3, 4, or 5 Infusion Reaction | 0 | 0

4. Primary Outcome: Severity of IRRs Following the Day 15 Infusion of Ocrelizumab in the Switching and the Comparator Groups Infusions
Description: The severity of IRRs will be assessed following each infusion of ocrelizumab in the switching and comparator group using the National Cancer Institute's Common Terminology for Adverse Events Scale (Grades range from 1-5, with higher Grades indicating more severe reactions). The frequency of each severity grade of IRR will be compared in a similar fashion.
Time Frame: Day 15, pre-study infusions
Population: The Switching group received 3 infusions (Day 1, Day 15 and week 24), and the Comparator group received 2 infusions. Proportion of IRRs are taken out of total number of infusions. This analysis is comparing IRRs of the Switching group's Day 15 infusion, with the comparator group's pre-study infusion 1 and 2.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Switching Group | Comparator Group
Number analyzed (Participants) | 100 | 100
Number analyzed (Infusions) | 100 | 200
Infusions
  No Infusion Reaction | 96 | 172
  Grade 1 Infusion Reaction | 0 | 3
  Grade 2 Infusion Reaction | 4 | 25
  Grade 3, 4, and 5 Infusion Reaction | 0 | 0

5. Primary Outcome: Severity of IRRs Following the Week 24 Infusion of Ocrelizumab in the Switching and the Comparator Groups Infusions
Description: as for outcome 3
Time Frame: Week 24, pre-study infusions
Population: The Switching group received 3 infusions (Day 1, Day 15 and week 24), and the Comparator group received 2 infusions. Proportion of IRRs are taken out of total number of infusions. This analysis is comparing IRRs of the Switching group's Week 24 infusion, with the comparator group's pre-study infusion 1 and 2.
Measure: Number; unit: Infusions
Units Other Than Participants: Infusions
Arm/Group | Switching Group | Comparator Group
Number analyzed (Participants) | 100 | 100
Number analyzed (Infusions) | 100 | 200
Infusions
  No Infusion Reaction | 88 | 172
  Grade 1 Infusion Reaction | 9 | 3
  Grade 2 Infusion Reaction | 3 | 25
  Grade 3, 4, and 5 Infusion Reaction | 0 | 0

6. Primary Outcome: Proportion of Patients With an IRR at Day 1 Versus Day 15 and Week 24 Infusions
Description: We will also compare the proportion of patients with an IRR following day 1 infusion versus the proportion of patients with an IRR at day 15 and month 6 infusions of ocrelizumab in the switching group.
Time Frame: Day 1, Day 15, Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Switching Group - Day 1 Infusion; Switching Group - Day 15 Infusion; Switching Group - Week 24 Infusion: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
Arm/Group | Switching Group - Day 1 Infusion | Switching Group - Day 15 Infusion | Switching Group - Week 24 Infusion
Number analyzed (Participants) | 100 | 100 | 100
Participants | 14 | 4 | 12
Statistical Analysis 1: Comparison: Switching Group - Day 1 Infusion vs Switching Group - Day 15 Infusion; Test type: Superiority; p = 0.0075, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = .2857, 95% CI 2-sided [.1072 to .7613]
Statistical Analysis 2: Comparison: Switching Group - Day 1 Infusion vs Switching Group - Week 24 Infusion; Test type: Superiority; p = 0.5930, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = .8571, 95% CI 2-sided [.4868 to 1.5093]
Statistical Analysis 3: Comparison: Switching Group - Day 15 Infusion vs Switching Group - Week 24 Infusion; Test type: Superiority; p = 0.0209, Generalized estimating equations; GEE was used because there are repeated measures on subjects; Risk Ratio (RR) = 3.0000, 95% CI 2-sided [1.1260 to 7.9932]

7. Secondary Outcome: Presence of Ocrelizumab Anti-drug Anti-bodies
Description: Proportion of ocrelizumab patients who test positive for ocrelizumab anti-drug anti-bodies
Time Frame: Day 1 and Week 24
Population: Reporting proportions of patients. 95% confidence intervals calculating using either the standard Z score method or the exact Clopper-Pearson method as necessary.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Switching Group - Day 1 Infusion | Switching Group - Week 24 Infusion
Number analyzed (Participants) | 100 | 100
percentage of patients | 1.00 [0.03 to 5.45] | 1.00 [0.03 to 5.45]

8. Secondary Outcome: Presence of Rituximab Anti-drug Anti-bodies
Description: Proportion of patients who test positive for rituximab anti-drug anti-bodies.
Time Frame: Day 1 and Week 24
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Switching Group - Day 1; Switching Group - Week 24: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
Arm/Group | Switching Group - Day 1 | Switching Group - Week 24
Number analyzed (Participants) | 100 | 100
percentage of patients | 16.00 [8.81 to 23.19] | 7.00 [2.86 to 13.89]

9. Secondary Outcome: B Cell Depletion (CD19)
Description: Proportion of patients with CD19% <= 1%.
Time Frame: Day 1, Week 24, 1 Year
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Switching Group - 1 Year: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
Arm/Group | Switching Group - Day 1 | Switching Group - Week 24 | Switching Group - 1 Year
Number analyzed (Participants) | 98 | 100 | 93
percentage of patients | 57.14 [47.35 to 66.94] | 92.00 [84.84 to 96.48] | 90.32 [82.42 to 95.48]

10. Secondary Outcome: B Cell Depletion (CD20)
Description: Proportion of patients with CD20% <= 1%
Time Frame: Day 1, Week 24, 1 Year
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Switching Group - Day 1 | Switching Group - Week 24 | Switching Group - 1 Year
Number analyzed (Participants) | 97 | 100 | 88
percentage of patients | 56.70 [46.84 to 66.56] | 92.00 [84.84 to 96.48] | 88.64 [82.01 to 95.27]

11. Secondary Outcome: Cytokine: Eotaxin - Pre-Post Infusion - Day 1
Description: Comparing Eotaxin concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: Change in mean concentration between pre and post infusion. Only cytokines with statistically significant pre-post changes reported.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Switching Group - Day 1 - Pre Infusion: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
  Pre-Infusion
- Switching Group - Day 1 - Post Infusion: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
  Post-Infusion
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 117.44 (50.19) | 101.41 (55.94)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.005, t-test, 2 sided — Controlled for the false discovery rate (alpha = 0.05) for all cytokines on day 1 using the Benjamini-Hochberg procedure; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = --16.03, 95% CI 2-sided [-27.05 to -5.01] — Mean of post minus pre

12. Secondary Outcome: Cytokine: IFN-gamma - Pre-Post Infusion - Day 1
Description: Comparing IFN-gamma concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 2.03 (1.42) | 4.58 (5.28)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 2.55, 95% CI 2-sided [1.54 to 3.56] — Mean of post minus pre

13. Secondary Outcome: Cytokine: IL-10 - Pre-Post Infusion - Day 1
Description: Comparing IL-10 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 0.18 (0.27) | 8.75 (11.28)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Median Difference (Net) = 8.58, 95% CI 2-sided [6.33 to 10.82] — Mean of post minus pre

14. Secondary Outcome: Cytokine: IL-12/IL-23p40 - Pre-Post Infusion - Day 1
Description: Comparing IL-12/IL-23p40 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 59.79 (38.79) | 52.42 (35.11)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = -7.37, 95% CI 2-sided [-10.19 to -4.55] — Mean of post minus pre

15. Secondary Outcome: Cytokine: IL-16 - Pre-Post Infusion - Day 1
Description: Comparing IL-16 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 85.48 (40.77) | 129.80 (80.10)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 44.32, 95% CI 2-sided [29.59 to 59.05] — Mean of post minus pre

16. Secondary Outcome: Cytokine: IL-1RA - Pre-Post Infusion - Day 1
Description: Comparing IL-1RA concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 196.71 (202.10) | 550.06 (920.23)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0002, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 353.35, 95% CI 2-sided [175.23 to 531.46] — Mean of post minus pre

17. Secondary Outcome: Cytokine: IL-27 - Pre-Post Infusion - Day 1
Description: Comparing IL-27 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 643.32 (269.50) | 820.23 (340.37)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 176.90, 95% CI 2-sided [124.50 to 229.31] — Mean of post minus pre

18. Secondary Outcome: Cytokine: IL-6 - Pre-Post Infusion - Day 1
Description: Comparing IL-6 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 0.29 (0.29) | 0.49 (0.56)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0020, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 0.19, 95% CI 2-sided [0.07 to 0.32] — Mean of post minus pre

19. Secondary Outcome: Cytokine: IL-7 - Pre-Post Infusion - Day 1
Description: Comparing IL-7 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 0.84 (0.36) | 1.38 (2.98)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 0.55, 95% CI 2-sided [0.32 to 0.77] — Mean of post minus pre

20. Secondary Outcome: Cytokine: IL-8(HA) - Pre-Post Infusion - Day 1
Description: Comparing IL-8(HA) concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 306.89 (186.64) | 260.73 (147.40)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0091, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = -46.16, 95% CI 2-sided [-80.61 to -11.72] — Mean of post minus pre

21. Secondary Outcome: Cytokine: MCP-1 - Pre-Post Infusion - Day 1
Description: Comparing MCP-1 concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 34.83 (14.37) | 90.09 (146.18)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0002, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 55.26, 95% CI 2-sided [27.00 to 83.52] — Mean of post minus pre

22. Secondary Outcome: Cytokine: MDC - Pre-Post Infusion - Day 1
Description: Comparing MDC concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 468.96 (138.66) | 451.72 (139.53)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0044, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = -17.24, 95% CI 2-sided [-28.96 to -5.51] — Mean of post minus pre

23. Secondary Outcome: Cytokine: MIP-1alpha - Pre-Post Infusion - Day 1
Description: Comparing MIP-1alpha concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 29.50 (26.72) | 45.52 (34.45)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 16.01, 95% CI 2-sided [9.75 to 22.28] — Mean of post minus pre

24. Secondary Outcome: Cytokine: MIP-1beta - Pre-Post Infusion - Day 1
Description: Comparing MIP-1beta concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 24.27 (9.63) | 453.35 (671.64)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 429.08, 95% CI 2-sided [296.07 to 562.10] — Mean of post minus pre

25. Secondary Outcome: Cytokine: MIP-3alpha - Pre-Post Infusion - Day 1
Description: Comparing MIP-3alpha concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 3.90 (2.64) | 5.13 (5.70)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0101, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 1.23, 95% CI 2-sided [0.30 to 2.16] — Mean of post minus pre

26. Secondary Outcome: Cytokine: TARC - Pre-Post Infusion - Day 1
Description: Comparing TARC concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 24.02 (13.54) | 32.72 (21.79)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 8.69, 95% CI 2-sided [4.87 to 12.52] — Mean of post minus pre

27. Secondary Outcome: Cytokine: TNF-alpha - Pre-Post Infusion - Day 1
Description: Comparing TNF-alpha concentration between pre and post ocrelizumab infusion - Day 1
Time Frame: Day 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 1 - Pre Infusion | Switching Group - Day 1 - Post Infusion
Number analyzed (Participants) | 100 | 100
pg/ml | 0.99 (0.39) | 2.53 (2.64)
Statistical Analysis 1: Comparison: Switching Group - Day 1 - Pre Infusion vs Switching Group - Day 1 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 11, analysis 1]; Paired T-test. Degrees of freedom = 99; Mean Difference (Net) = 1.53, 95% CI 2-sided [1.04 to 2.03] — Mean of post minus pre

28. Secondary Outcome: Cytokine: Exotaxin - Pre-Post Infusion - Day 15
Description: Comparing Exotaxin concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Switching Group - Day 15 - Pre Infusion: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
  Pre-Infusion
- Switching Group - Day 15 - Post Infusion: 600 mg of ocrelizumab will be administered as one 600-mg IV infusions at a scheduled interval of every 24 weeks. The first dose of ocrelizumab will be a split dose of 300 mg on day 1 and day 15 followed by 600 mg, six months later. Each ocrelizumab infusion should be given as a slow IV infusion over approximately 150 minutes (2.5 hours) for the 300-mg dose. Ocrelizumab must not be administered as an IV push or bolus. Well-adjusted infusion pumps should be used to control the infusion rate, and ocrelizumab should be infused through a dedicated line.
  Ocrelizumab: A humanized monoclonal antibody that targets CD20 and selectively depleted CD-20 expressing B cells
  Post-Infusion
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 128.38 (54.32) | 95.79 (60.29)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — 99 patients with non-missing change scores used. Controlled for the false discovery rate (alpha = 0.05) for all cytokines on day 15 using the Benjamini-Hochberg procedure; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -33.17, 95% CI 2-sided [-38.91 to -27.44] — Mean of post minus pre. 99 usable change scores

29. Secondary Outcome: Cytokine: IFN-gamma - Pre-Post Infusion - Day 15
Description: Comparing IFN-gamma concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 2.02 (1.37) | 1.40 (1.49)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0008, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -0.62, 95% CI 2-sided [-0.98 to -0.26] — Mean of post minus pre. 99 usable change scores

30. Secondary Outcome: Cytokine: IL-10 - Pre-Post Infusion - Day 15
Description: Comparing IL-10 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 0.12 (0.12) | 2.12 (3.91)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = 2.01, 95% CI 2-sided [1.23 to 2.79] — Mean of post minus pre. 99 usable change scores

31. Secondary Outcome: Cytokine: IL-12/IL-23p40 - Pre-Post Infusion - Day 15
Description: Comparing IL-12/IL-23p40 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 49.36 (31.75) | 41.31 (29.24)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -7.84, 95% CI 2-sided [-9.87 to -5.81] — Mean of post minus pre. 99 usable change scores

32. Secondary Outcome: Cytokine: IL-16 - Pre-Post Infusion - Day 15
Description: Comparing IL-16 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 90.35 (54.78) | 76.62 (29.78)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0022, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -14.20, 95% CI 2-sided [-23.15 to -5.25] — Mean of post minus pre. 99 usable change scores

33. Secondary Outcome: Cytokine: IL-1beta - Pre-Post Infusion - Day 15
Description: Comparing IL-1beta concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 0.65 (0.73) | 0.95 (0.72)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = 0.30, 95% CI 2-sided [0.17 to 0.43] — Mean of post minus pre. 99 usable change scores

34. Secondary Outcome: Cytokine: IL-7 - Pre-Post Infusion - Day 15
Description: Comparing IL-7 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 0.88 (0.64) | 1.29 (0.95)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = 0.41, 95% CI 2-sided [0.22 to 0.61] — Mean of post minus pre. 99 usable change scores

35. Secondary Outcome: Cytokine: IL-8 - Pre-Post Infusion - Day 15
Description: Comparing IL-8 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 1.82 (1.48) | 1.09 (0.80)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -0.72, 95% CI 2-sided [-0.95 to -0.50] — Mean of post minus pre. 99 usable change scores

36. Secondary Outcome: Cytokine: MCP-1 - Pre-Post Infusion - Day 15
Description: Comparing MCP-1 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 35.57 (18.08) | 16.33 (9.24)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -19.31, 95% CI 2-sided [-22.64 to -15.98] — Mean of post minus pre. 99 usable change scores

37. Secondary Outcome: Cytokine: MCP-4 - Pre-Post Infusion - Day 15
Description: Comparing MCP-4 concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 37.38 (23.70) | 30.38 (15.08)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -6.96, 95% CI 2-sided [-9.85 to -4.08] — Mean of post minus pre. 99 usable change scores

38. Secondary Outcome: Cytokine: MDC - Pre-Post Infusion - Day 15
Description: Comparing MDC concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 458.13 (154.72) | 435.00 (165.94)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0061, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -23.22, 95% CI 2-sided [-39.66 to -6.78] — Mean of post minus pre. 99 usable change scores

39. Secondary Outcome: Cytokine: MIP-1beta - Pre-Post Infusion - Day 15
Description: Comparing MIP-1beta concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 23.09 (9.46) | 17.23 (7.80)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -5.69, 95% CI 2-sided [-7.24 to -4.14] — Mean of post minus pre. 99 usable change scores

40. Secondary Outcome: Cytokine: MIP-3alpha - Pre-Post Infusion - Day 15
Description: Comparing MIP-3alpha concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 4.15 (4.32) | 3.31 (2.83)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p = 0.0077, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.45 to -0.23] — Mean of post minus pre. 99 usable change scores

41. Secondary Outcome: Cytokine: TNF-alpha - Pre-Post Infusion - Day 15
Description: Comparing TNF-alpha concentration between pre and post ocrelizumab infusion - Day 15
Time Frame: Day 15
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Switching Group - Day 15 - Pre Infusion | Switching Group - Day 15 - Post Infusion
Number analyzed (Participants) | 100 | 99
pg/ml | 1.14 (0.45) | 0.81 (0.34)
Statistical Analysis 1: Comparison: Switching Group - Day 15 - Pre Infusion vs Switching Group - Day 15 - Post Infusion; Paired T-test for change in means. Null hypothesis: no pre-post difference; Test type: Other; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 28, analysis 1]; Paired T-test. Degrees of freedom = 98; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.37 to -0.27] — Mean of post minus pre. 99 usable change scores

ADVERSE EVENTS:
Time Frame: 1 year - enrollment to month 12 infusion.
Description: Because data for the comparator group was collected retrospectively using chart review, 0 participants in that group were at risk for All-Cause Mortality, and All-Cause Mortality was not monitored for that group.
Arm/Group | Switching Group | Comparator Group
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/0
Serious Adverse Events (participants affected / at risk) | 8/100 | 0/100
Other Adverse Events (participants affected / at risk) | 52/100 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching Group (N=100) | Comparator Group (N=100)
clostridium difficile colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Immune system disorders) | 1 (1) | 0 (0)
Hip Dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Unknown pulmonary complications (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Liver and renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Encephalopathy (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switching Group (N=100) | Comparator Group (N=100)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 36 (47) | 0 (0)
Headache (General disorders) | 14 (17) | 0 (0)
Nausea (General disorders) | 14 (14) | 0 (0)
Numbness (General disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02980042/Prot_SAP_000.pdf